CLINICAL TRIAL: NCT04055948
Title: Building Family Caregiver Skills Using a Simulation-Based Intervention for Care of Patients With Cancer
Brief Title: Building Family Caregiver Skills Using a Simulation-Based Intervention for Care of Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE4Y19; 1R37CA240707-01 (NIH)
Record Dates: First submitted 2019-08-07; First posted 2019-08-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Patient and family caregiver dyads are enrolled in this 2-group, prospective, randomized controlled design to test the effect of a caregiver intervention during radiation therapy.
  The study enrolled a total of 242 dyads(484 participants)
Who Masked: Investigator
Masking Description: Research Assistant (RA) will be blind to which group CG is assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard of Care (No Intervention): CG(caregivers)/CP(cancer patients) dyads
  - All participants will be screened for health literacy using a 4-item Brief Health Literacy Screening Tool (BRIEF)
- Intervention (Experimental): CG/CP dyads
  * All participants will be screened for health literacy using a 4-item Brief Health Literacy Screening Tool (BRIEF)
  * Three in-person, one-on-one teaching sessions with the caregiver during radiation treatments, followed by a telephone booster contact 2 weeks post-treatment.
  Interventions: Behavioral: One-on-one teaching sessions; Behavioral: Telephone booster contact

INTERVENTIONS:
Behavioral: One-on-one teaching sessions — One-on-one teaching sessions with the caregiver during radiation treatments. (note - intervention sessions 2 & 3 delivered by phone during COVID-19)
  Arms: Intervention
Behavioral: Telephone booster contact — Telephone booster contact 2 weeks post-treatment.
  Arms: Intervention

SUMMARY:
The purpose of this study is to learn whether an education and support program can help caregivers feel more confident in technical and communication skills needed to care for a person with cancer. Patients with cancer and their caregivers face many challenges. These include learning about cancer and its treatment, coping with symptoms from illness and treatment side effects, making adjustments to usual activities, and managing the emotional effects of having a serious illness. This study is testing whether different forms of education and support can help caregivers feel better prepared. To find out if education about caregiving and different kinds of support are effective, study personnel will compare approaches to help find ways to improve the services that are provided to caregivers during cancer treatment. About 180 patients and their caregivers at the Seidman Cancer Center will take part in this study. Participating in research is voluntary and this study is funded by the National Institute of Health.

DETAILED DESCRIPTION:
This is a 2-group, prospective, randomized controlled design to test the effect of an intervention, as compared to a usual care control group, on family caregivers (CG) outcomes, patient outcomes, and healthcare utilization outcomes during treatment.

The objectives of this study are to:

* Evaluate the effect of a CG intervention, as compared to a control group, on CG primary (anxiety) and secondary (depression, health-related quality of life [HRQOL], and fatigue) outcomes.
* Measure the effect of the intervention, as compared to a control group, on patient outcomes (HRQOL and interrupted treatment course), and healthcare utilization outcomes (unplanned hospital admissions, unplanned emergency room visits, and unplanned use of intravenous [IV] fluids).
* Determine if CG self-efficacy mediates the effect of the intervention on CG anxiety.
* Determine if patient illness factors, care demands (hours per week spent caregiving), and patient and CG demographic factors moderate the relationship between the intervention and CG outcomes.
* Compare the costs of healthcare utilization (unplanned hospital admission, unplanned emergency room visits, and unplanned use of IV fluids) between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria (for patients):

* Diagnosis of stage I, II, III cancers of the rectum, anus, and esophagus; stage III NSCLC; and stage I - IV A/B head/neck (tongue, gum, oral cavity, nasopharynx, oropharynx, hypopharynx, parotid, or larynx).
* Receiving their first course of radiation therapy.
* Has an identified family CG who is willing to participate.

Inclusion Criteria (for CGs):

* Family member or friend of an adult patient described above; and
* Identified by the patient as his/her primary CG, who is providing daily assistance and/or emotional support.

Exclusion Criteria:

* Patients who do not have a caregiver will be excluded.
* CGs of patients who are receiving hospice care will be excluded because of the patient's poor prognosis and multiple issues associated with end-of-life care.
* CGs who are themselves undergoing active cancer treatment will be excluded (hormonal treatment allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
CG anxiety at 20 weeks post-treatment | 20 weeks post treatment
  Difference in CG anxiety between the intervention and control groups at 20 weeks post-radiation treatment.
  CG anxiety will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form 7a. This 7-item questionnaire assesses self-reported fear, worry, anxiety, tension, nervousness, and restlessness in the family caregiver over the last 7 days.
  This outcome will be reporting the average T-score for anxiety as measured by the PROMIS scale. Raw scores range from 7 to 35. Each participant's raw score on the scale will be converted to a standardized T-score that has a mean of 50 and a standard deviation of 10. A higher T-score represents greater anxiety. For example, a T-score of 60 is one standard deviation worse anxiety than average.

SECONDARY OUTCOMES:
CG anxiety at the end of radiation treatment | At end of treatment, average of seven weeks
  Difference in CG anxiety between the intervention and control groups at the end of radiation treatment
  CG anxiety will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form 7a. This 7-item questionnaire assesses self-reported fear, worry, anxiety, tension, nervousness, and restlessness in the family caregiver over the last 7 days.
  This outcome will be reporting the average T-score for anxiety as measured by the PROMIS scale. Raw scores range from 7 to 35. Each participant's raw score on the scale will be converted to a standardized T-score that has a mean of 50 and a standard deviation of 10. A higher T-score represents greater anxiety. For example, a T-score of 60 is one standard deviation worse anxiety than average.
CG anxiety at 4 weeks post treatment | 4 weeks post treatment
  CG anxiety between the intervention and control groups at 4 weeks post treatment.
  CG anxiety will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form 7a. This 7-item questionnaire assesses self-reported fear, worry, anxiety, tension, nervousness, and restlessness in the family caregiver over the last 7 days.
  This outcome will be reporting the average T-score for anxiety as measured by the PROMIS scale. Raw scores range from 7 to 35. Each participant's raw score on the scale will be converted to a standardized T-score that has a mean of 50 and a standard deviation of 10. A higher T-score represents greater anxiety. For example, a T-score of 60 is one standard deviation worse anxiety than average.
CG depression | at baseline, at end of treatment (average of seven weeks), and at 4 and 20 weeks post treatment
  CG depression will be measured with the PROMIS Depression Short Form 8b. This 8-item questionnaire assesses caregiver self-reported negative mood (sadness, guilt), views of self (worthlessness), and social cognition (loneliness), as well as decreased positive affect and engagement. It assesses depression over the last 7 days.
  This outcome will be reporting the average T-score for depression as measured by the PROMIS scale. Raw scores range from 8 to 40. Each participant's raw score on the scale will be converted to a standardized T-score that has a mean of 50 and a standard deviation of 10. A higher T-score represents greater depression. For example, a T-score of 60 is one standard deviation worse depression than average.
CG HRQOL as measured by PROMIS Global Health Scale Global Physical Health and Global Mental Health domains | at baseline, at end of treatment (average of seven weeks), and at 4 and 20 weeks post treatment
  The PROMIS Global Health Scale will be scored as two separate domains - Global Physical Health and Global Mental Health. These domains are not combined for a total score. Raw scores range from 4 to 20. Each participant's raw score on the scale will be converted to a standardized T-score that has a mean of 50 and a standard deviation of 10. A higher T-score represents better health (Global Physical Health or Global Mental Health) than the general population. For example, a T-score of 60 is one standard deviation better health than average
CG fatigue | at baseline, at end of treatment (average of seven weeks), and at 4 and 20 weeks post treatment
  CG fatigue will be measured with the PROMIS Fatigue Short Form 7a, a 7-item questionnaire that evaluates the self-reported experience of fatigue (frequency, duration, intensity) and the impact of fatigue on daily activities. It assesses fatigue over the last 7 days.
  This outcome will be reporting the average T-score for fatigue. Raw scores range from 7 to 35. Each participant's raw score on the scale will be converted to a standardized T-score that has a mean of 50 and a standard deviation of 10. A higher T-score represents greater fatigue. For example, a T-score of 60 is one standard deviation worse fatigue than average.
Participant HRQOL (cancer patient) as measured by FACT-C | at baseline, at end of treatment (average of seven weeks), and at 4 and 20 weeks post treatment
  Participant HRQOL will be measured using the disease-specific versions of FACT-G that include common subscales (physical, social, emotional, and functional well-being) plus cancer-specific questions. The effect of the intervention on HRQOL across diagnoses will be analyzed using the common subscales. The symptom experience with each diagnostic group will be described using the cancer-specific subscale.
  Participants rate their response to each item on a 5-point Likert-type scale. After reverse-scoring negatively worded questions, items are summed. Higher scores indicate better quality of life.
  The FACT - Colorectal (FACT-C, Version 4) is a 37-item questionnaire that measures self-reported HRQOL in patients with colorectal cancer over the last 7 days.
Participant HRQOL (cancer patient) as measured by FACT-H&N | at baseline, at end of treatment (average of seven weeks), and at 4 and 20 weeks post treatment
  Participant HRQOL will be measured using the disease-specific versions of FACT-G that include common subscales (physical, social, emotional, and functional well-being) plus cancer-specific questions. The effect of the intervention on HRQOL across diagnoses will be analyzed using the common subscales. The symptom experience with each diagnostic group will be described using the cancer-specific subscale.
  Participants rate their response to each item on a 5-point Likert-type scale. After reverse-scoring negatively worded questions, items are summed. Higher scores indicate better quality of life.
  The FACT - Head & Neck Scale (FACT-H&N, Version 4) is a 39-item questionnaire that assesses self-reported HRQOL in patients with head & neck cancer over the last 7 days
Participant HRQOL (cancer patient) as measured by FACT - E | at baseline, at end of treatment (average of seven weeks), and at 4 and 20 weeks post treatment
  Participant HRQOL will be measured using the disease-specific versions of FACT-G that include common subscales (physical, social, emotional, and functional well-being) plus cancer-specific questions. The effect of the intervention on HRQOL across diagnoses will be analyzed using the common subscales and will describe the symptom experience within each diagnostic group using the cancer-specific subscale.
  Participants rate their response to each item on a 5-point Likert-type scale. After reverse-scoring negatively worded questions, items are summed. Higher scores indicate better quality of life.
  The FACT - Esophageal (FACT-E)
Participant HRQOL (cancer patient) as measured by FACT-L | at baseline, at end of treatment (average of seven weeks), and at 4 and 20 weeks post treatment
  Participant HRQOL will be measured using the disease-specific versions of FACT-G that include common subscales (physical, social, emotional, and functional well-being) plus cancer-specific questions. The effect of the intervention on HRQOL across diagnoses will be analyzed using the common subscales and will describe the symptom experience within each diagnostic group using the cancer-specific subscale.
  Participants rate their response to each item on a 5-point Likert-type scale. After reverse-scoring negatively worded questions, items are summed. Higher scores indicate better quality of life.
  The FACT - Lung (FACT-L)
Interrupted treatment | At end of treatment, average of seven weeks
  Interrupted Radiation Treatment Course, defined as the total number of missed treatment days due to patient or caregiver reasons, will be determined from the patient's radiation therapy treatment record. Number of days of each episode of absence from treatment will also be recorded.
Healthcare utilization cost | at baseline, at end of treatment (average of seven weeks), and at 4 and 20 weeks post treatment
  Healthcare utilization includes unplanned hospital admission, unplanned emergency room visits, and unplanned IV fluid use for treatment of dehydration.
  These variables will be combined to compute a "healthcare utilization cost" for each participant. Medicare reimbursement rates will be used to estimate costs regardless of the age or insurance of the participant. Using the DRG, diagnosis and procedure codes we will determine what Medicare "would have paid" for those services, and will use that as a proxy for cost. Cost of IV fluids will be estimated using wholesale acquisition cost. Mean differences between the intervention and control groups will be analyzed using a two sample t-test for independent means.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mazanec, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

REFERENCES:
- [Derived] Park S, Blackstone EC, Mazanec SR. Exploring the determinants of health literacy and its effects on health-related outcomes in family caregivers of patients with cancer. Support Care Cancer. 2025 Apr 29;33(5):433. doi: 10.1007/s00520-025-09494-7. PMID 40299112
- [Derived] Mazanec SR, Blackstone E, Daly BJ. Building family caregiver skills using a simulation-based intervention for care of patients with cancer: protocol for a randomized controlled trial. BMC Nurs. 2021 Jun 9;20(1):93. doi: 10.1186/s12912-021-00612-4. PMID 34107914